CLINICAL TRIAL: NCT00192907
Title: Inflammation and Infection in Trauma, Role in Posttraumatic Complications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: KF 01-160/02 Main
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the relationship between trauma, the immune system, biochemical changes in the first 24 h and subsequent complications and mortality

DETAILED DESCRIPTION:
The immune system plays a role in the development of complications after severe trauma, but we do not know how. Equally, biochemical changes measured in the blood after trauma (eg. bloodglucose, GC-globulin, coagulation parameters etc.) may predict the prognosis and the degree of complcations. Two significant complications are infection and organ failure, which may prolong hospitalisation and increase mortality.

In the study we collected samples from blood and body surfaces to determine changes in cytokines, biochemistry, bacterial flora, and subsequent complications. We compare the changes in between groups of the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of multiple trauma
* Age >/= 18 years
* Direct referral from scene of accident

Exclusion Criteria:

* Major burn injury
* HIV positiv
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2003-03; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stensballe, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Dk-2100 Copenhagen, Denmark

REFERENCES:
- [Derived] Johansson PI, Stensballe J, Rasmussen LS, Ostrowski SR. A high admission syndecan-1 level, a marker of endothelial glycocalyx degradation, is associated with inflammation, protein C depletion, fibrinolysis, and increased mortality in trauma patients. Ann Surg. 2011 Aug;254(2):194-200. doi: 10.1097/SLA.0b013e318226113d. PMID 21772125